CLINICAL TRIAL: NCT01367821
Title: Quorum Sensing Signal Molecules (QSSMs) and Immune Dysfunction in Patients Undergoing Endoscopic Retrograde Cholangiopancreatography (ERCP) for Obstructive Jaundice
Brief Title: Immune Function in Patients With Obstructive Jaundice
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 10040; 10/H0408/53 (Other: Nottingham Research Ethics Committee 2)
Record Dates: First submitted 2011-05-31; First posted 2011-06-07 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Obstructive Jaundice; Disease as Reason for ERCP; Immune Dysfunction; Immune Tolerance
Keywords: Obstructive jaundice; ERCP; Immune dysfunction; Endotoxin tolerance; Quorum sensing
MeSH Terms: conditions — Jaundice, Obstructive; Immune System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma Bile
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with obstructive jaundice: Patients with obstructive jaundice
- Healthy volunteers: Healthy volunteers

SUMMARY:
Patients with obstructive jaundice (OJ) often require surgical, endoscopic or radiological interventions to facilitate biliary drainage and relieve jaundice. However it is known that patients with OJ have increased surgical risks than non-jaundiced patients undergoing the same procedures. Surgery for severe OJ is associated with a significant post-operative mortality (10-15%) and morbidity (30-65%). The commonest complications are related to sepsis but the pathophysiological mechanisms behind this susceptibility to bacterial infection are not clear. Recent work has shown a pivotal role of bile in the maintenance of enterocyte tight junctions and the expression of tight junction-associated proteins which could account for the translocation of enteric bacteria and bacterial products to mesenteric lymph node complexes, the portal circulation and subsequently the liver. Some of these bacterial products, such as endotoxin and quorum sensing signalling molecules (QSSMs), have immunomodulatory properties which may dampen normal immune responses to infection resulting in life-threatening organ dysfunction. Bacterial endotoxin and quorum sensing signalling molecules (QSSMs) represent good candidates for the mediators of this immune suppression and although there is a compelling case for their involvement in the pathogenesis of sepsis, evidence to support their involvement in the aetiology of infection in OJ is currently lacking.

DETAILED DESCRIPTION:
Obstructive jaundice (OJ) is a condition where a blockage of flow of bile from the liver leads to the accumulation of bile products in the blood resulting in yellowing and itching of the skin. Common causes of OJ include gallstones and also tumours of the pancreas or bile duct. Relieving this type of jaundice and treating the underlying cause can include endoscopic or surgical procedures. It is known however, that patients with OJ have increased surgical risks than non-jaundiced patients who undergo the same operations. Studies have shown that surgery for severe OJ is associated with a postoperative mortality in the region of 10-15% and morbidity rates of 30-65%. Complications related to bacterial infection are common and patients developing severe infections may require treatment with broad spectrum antibiotics with care in intensive or high dependency units.

Although antibiotics have proved invaluable in treating postoperative infections they carry the potential for adverse effects. Antibiotics can suppress normal gut bacteria and allow disease causing bacteria to proliferate, such as Clostridium difficile. This usually manifests as mild-to-moderate diarrhoea but can occasionally cause life-threatening bowel inflammation. The widespread use of antibiotics is also central to the development of bacterial strains with antibiotic resistance. This clinical problem also has economic, political and environmental implications for the National Health Service. Adherence to measures of infection control, education and antibiotic policy can minimise antibiotic resistance; however the limits surrounding such approaches have led to a demand for novel or alternative strategies.

It has recently been discovered that bacteria are able to communicate by producing specialised molecules known as quorum sensing signalling molecules (QSSMs). An accumulation of QSSMs in their surrounding environment allow for the bacteria to quantify the size of colonies. At specific colony sizes the concentration of QSSMs reaches a critical threshold leading to the activation of genes that cause an infection. Disruption of quorum sensing has been shown to reduce the severity of infection in animal studies and this has led to the development of inhibitors of quorum sensing as a possible strategy in antibacterial therapy.

Previous work conducted at the University of Nottingham has demonstrated that QSSMs also influence the number and function of a specific type of immune cell known as 'antigen presenting cells'. These cells are pivotal in allowing the immune system to recognise components of bacteria as foreign and thereby mount the appropriate response. It was found that large numbers of these types of cells underwent programmed cell death (cell suicide) in the presence of QSSMs compared to when QSSMs were absent. This mirrors the situation in blood sampled from patients with severe infections where there is a greater proportion of cell deaths among antigen presenting cells than other types of immune cell.

It is likely that the susceptibility to infectious complications in patients with obstructive jaundice is due to the interplay of various factors. The absence of intestinal bile has implications for the integrity of the bowel wall as a barrier, changes in gut microflora flora and translocation of both bacteria and their products. In addition, it is clear that a form of immune dysfunction occurs, which dampens the normal response following exposure to bacterial products. This immune dysfunction may avert powerful inflammatory cascades resulting in life-threatening multi organ dysfunction but at the expense of conditions that favour bacterial survival. QSSMs represent good candidates for the mediators of this immune dysfunction and although there is a compelling case for their involvement in the pathogenesis of sepsis, definitive evidence to support their role in infective processes in OJ is currently lacking.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive jaundice
* Willing to participate and able to give informed consent
* Alcohol abstinence during study

Exclusion Criteria:

* Acute Physiology and Chronic Health Evaluation (APACHE) II Score ≥8
* Severe neutropaenia
* Smokers/substance abuse
* Diabetes Mellitus
* Oral/IV Steroids
* On regular antibiotics
* Patients with active cholangitis
* Patients who have a history liver transplantation or chronic liver disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred to tertiary hepatopancreaticobiliary centre for investigation of obstructive jaundice and Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Change in monocyte cytokine responses to endotoxin stimulation | Baseline (pre ERCP) and post ERCP days 1, 7, 14 and 30
  Evaluation of monocyte cytokine responses to endotoxin stimulation at specified time points

SECONDARY OUTCOMES:
Change in concentration of systemic quorum sensing signaling molecules | Baseline (pre ERCP) and post ERCP days 1, 7, 14 and 30
  Evaluation of the presence of quorum sensing signalling molecules in the systemic circulation at specified time points

CONTACTS AND LOCATIONS:
Overall Officials: Abeed H Chowdhury, MBChB MRCS, Principal Investigator — University of Nottingham
Locations (1):
- Queen's Medical Centre, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Background] Blamey SL, Fearon KC, Gilmour WH, Osborne DH, Carter DC. Prediction of risk in biliary surgery. Br J Surg. 1983 Sep;70(9):535-8. doi: 10.1002/bjs.1800700910. PMID 6616158
- [Background] Han XC, Li JL, Han G. Surgical mortality in patients with malignant obstructive jaundice: a multivariate discriminant analysis. Hepatobiliary Pancreat Dis Int. 2003 Aug;2(3):435-40. PMID 14599955
- [Background] Povoski SP, Karpeh MS Jr, Conlon KC, Blumgart LH, Brennan MF. Association of preoperative biliary drainage with postoperative outcome following pancreaticoduodenectomy. Ann Surg. 1999 Aug;230(2):131-42. doi: 10.1097/00000658-199908000-00001. PMID 10450725
- [Background] Wang Q, Gurusamy KS, Lin H, Xie X, Wang C. Preoperative biliary drainage for obstructive jaundice. Cochrane Database Syst Rev. 2008 Jul 16;(3):CD005444. doi: 10.1002/14651858.CD005444.pub2. PMID 18677779
- [Background] Diggle SP, Crusz SA, Camara M. Quorum sensing. Curr Biol. 2007 Nov 6;17(21):R907-10. doi: 10.1016/j.cub.2007.08.045. No abstract available. PMID 17983563
- [Background] Martin CA, Hoven AD, Cook AM. Therapeutic frontiers: preventing and treating infectious diseases by inhibiting bacterial quorum sensing. Eur J Clin Microbiol Infect Dis. 2008 Aug;27(8):635-42. doi: 10.1007/s10096-008-0489-3. Epub 2008 Mar 6. PMID 18322716
- [Background] Williams P. Bacillus subtilis: a shocking message from a probiotic. Cell Host Microbe. 2007 Jun 14;1(4):248-9. doi: 10.1016/j.chom.2007.05.010. PMID 18005705
- [Background] Boontham P, Robins A, Chandran P, Pritchard D, Camara M, Williams P, Chuthapisith S, McKechnie A, Rowlands BJ, Eremin O. Significant immunomodulatory effects of Pseudomonas aeruginosa quorum-sensing signal molecules: possible link in human sepsis. Clin Sci (Lond). 2008 Dec;115(11):343-51. doi: 10.1042/CS20080018. PMID 18363571